CLINICAL TRIAL: NCT02622061
Title: A Clinical Investigation Determining the Discriminative Ability of the NIOX VERO NASAL to Differentiate Subjects With Primary Ciliary Dyskinesia From Healthy Controls
Brief Title: NIOX VERO Nasal Application in Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-051
Record Dates: First submitted 2015-12-01; First posted 2015-12-04 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: PCD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCD Subjects: Participants 5 and older with PCD.
- Healthy Subjects: Participants 5 and older without any pulmonary disease.

SUMMARY:
This is a multi-centre, single visit clinical investigation involving patients with known PCD vs. age matched healthy volunteers. This study involves 1 visit which will last one (1) to two (2) hours. Participants (and parent as applicable) will be asked for their consent to participate in the study. A brief medical history will be recorded, including information such as age, gender, height, weight, race, current medications and living environment. If the participant is a PCD patient, they will also be asked about their disease history. Prior to performing the nasal measurements, participants will receive instructions from study personnel and have the opportunity to practice. All participants will have a brief nasal exam and will also have to blow their nose before starting the measurements. Participants will be asked to perform nasal nitric oxide measurements using the tidal breathing method followed by the velum closed with expiration against resistance method.

The primary objective is to determine the feasibility and capability of the NIOX VERO to discriminate participants with PCD from those that are healthy. Information collected in this study will help researchers understand more about the diagnosis of and identification of patients with PCD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 5 years and older.
2. Anatomically, is able to complete the nasal NO measurements in both nostrils.
3. Cohort 1 - PCD Patients: Patients must have a confirmed diagnosis of PCD from one of the PCD diagnostic centres based on clinical phenotype PLUS diagnosis made by at least 1 of the following (the specifics about how diagnosis was made must be documented in their medical file):

   * A nasal biopsy or scraping showing a hallmark PCD defect such as, an outer (+/- inner) dynein arm defect, microtubule defect, or
   * A genetic test positive for bi-alleilic mutations in a known PCD-causing gene associated with the diagnosis of PCD (e.g., ARMC4, C21orf59, CCDC39, CCDC40, CCDC65, CCDC164, CCDC103, CCDC114, CCDC151, CCNO, DNAAF1 (LRRC50), DNAAF2 (KTU), DNAAF3, DNAH5, DNAH11, DNAI1, DNAI2, DNAL1, DYX1C1, HEATR2, HYDIN, LRRC6, MCIDAS, NME8 (TXNDC3), ODA/IDA, OFD1, RPGR, RSPH3, RSPH4A, RSPH9, SPAG1, ZMYND10), or
   * EU Centres Only: A low nasal NO (determined by a chemiluminescent analyser) plus either:

     * at least 2 separate occasions with 'hallmark' changes on high-speed video microscopy, or
     * demonstration of mislocalisation of ciliary proteins by immunofluorescence microscopy.
4. Cohort 2 - Healthy Patients: Healthy, non-atopic, non-smoking patients (defined as patient with no airway or immune problems, no recent significant injury, no systemic infection, no systemic inflammation, no allergies or asthma).

Exclusion Criteria:

1. Currently smokes or it has been less than 6 months from quitting.
2. Has had a nose bleed within the past 2 weeks.
3. Has acute respiratory symptoms or signs of an upper or lower respiratory tract infection.
4. Use of nasal medication as described below:

   * Xolair ≤180 days prior to nNO measurement
   * Oral or Systemic Corticosteroids ≤30 days prior to nNO measurement
   * Inhaled, nebulized, or intranasal corticosteroids ≤30 days prior to nNO measurement
   * Nasal or oral decongestants or antihistamines ≤14 days prior to nNO measurement
   * Leukotriene receptor antagonists ≤30 days prior to nNO measurement
5. Has an obstruction or anatomy that prevents a nasal measurement from being performed (as confirmed by simple visual inspection by the Investigator).
6. Has Cystic Fibrosis.
7. Has a documented primary or acquired immunodeficiency.
8. Is undergoing treatment with NO-releasing drugs (such as nitrates or molsidomine).
9. Has had food or beverage intake (other than water) or has participated in strenuous exercise within 1 hour of nasal NO measurement
10. Is unwilling or unable to provide consent to participate (self, parent or legal guardian).
11. PCD Patients Only: Has mutations with RSPH1 since nasal NO may not be low in these patients.
12. PCD Patients Only: Has not had a standard clinical evaluation to address other potential causes of chronic oto-sino- pulmonary disease.
13. Healthy Patients Only: Atopy or the presence of any of the following: a recent significant injury (i.e., within 1-2 weeks), systemic inflammation, airway or immune problem, asthma or allergies.
14. In the US only: Patients may not be related to a member of the Study Personnel.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a multi-center, single visit clinical investigation involving patients with known PCD [Cohort 1] vs. age matched healthy volunteers [Cohort 2].
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the analysis of the means of the successful nNO measurements in Subjects with PCD as compared with Healthy Subjects in the Evaluable Population. | After a single 1-2 hour visit

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Rickard, MD, Study Director — Aerocrine AB
Locations (5):
- United States (2):
  - St Louis, St Louis, Missouri
  - Chapel Hill, Chapel Hill, North Carolina
- Denmark, Copenhagen, Denmark
- Paris, Paris, France
- Germany, Münster, Germany

IPD SHARING:
Plan to Share IPD: No